CLINICAL TRIAL: NCT07210814
Title: Pilot Study on the Activity of Commercially Available Mouthwashes Againgst Entamoeba Spp.
Brief Title: Activity of Mouthwashes Againgst Entamoeba Spp.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Martina Koehsler, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1368/2025
Record Dates: First submitted 2025-09-11; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Parasite Infestation
Keywords: Entamoeba gingivalis; mouthwash
MeSH Terms: conditions — Parasitic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- regular participants (Experimental): inital sampling, plaque and saliva is collected by a medical professional, for 7 days a mouthwash is used twice dayly for 30 seconds, final sampling, plaque and saliva is collected by a medical professional
  Interventions: Procedure: saliva and plaque sample collection for analysis; Other: using commercial mouthwash

INTERVENTIONS:
Procedure: saliva and plaque sample collection for analysis — For collection of plaque two different gingival sites are selected for sampling in each participant. Prior to sampling, supragingival plaque is removed with a sterile instrument. Subgingival plaque is then collected from the same site using a sterile Gracey curette.
  Saliva samples are collected using a commercially available saliva collection kit (Sallivete®, SARSTEDT AG, Germany). Participants should open the Sallivete® tube, remove the synthetic swab, and place it in their mouth for 1-2 minutes, ensuring it moves around to facilitate optimal saliva collection while avoiding chewing.
Other: using commercial mouthwash — Participants use the commercial mouthwash octenident (cosmetic) twice daily after their normal dental routine for 30 seconds for consecutive seven days

SUMMARY:
The amoeba Entamoeba gingivalis colonizes the human oral cavity, where it can actively destroy tissue and cause local inflammation. Currently, there is no standard treatment for E. gingivalis infection. Even during treatment for periodontitis, there is no specific treatment targeting E. gingivalis, although this could significantly improve the effectiveness and long-term results of periodontitis therapy. Octenidine is an antiseptic agent used for disinfecting skin, mucous membranes, and wounds. It is effective against bacteria, fungi, and some viruses. octenident® is a commercially available cosmetic mouthwash containing octenidine as the active ingredient. Its efficacy against Entamoeba spp. will be tested in vitro. Because E. gingivalis is very difficult to cultivate under laboratory conditions, and in vitro testing may not be feasible, the effect of using the mouthwash octenident® (cosmetic product) twice daily for 30 seconds over a 7-day period on the quantity of E. gingivalis will be evaluated in healthy volunteers using quantitative real-time PCR, a technique enabling the comparison of E. gingivalis DNA before and after the use of octenident®.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Able and willing to provide written informed consent
* Positive identification of Entamoeba gingivalis in oral samples collected during screening, confirmed by specific PCR

Exclusion Criteria:

* Antibiotic therapy or periodontal treatment within the last 6 months
* Current orthodontic treatment
* Underlying systemic diseases (e.g., diabetes mellitus)
* Autoimmune diseases
* Acute infections and other conditions requiring medication
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in E. gingivalis DNA quantity after using the mouthwash octenident®. | 8 days, pre-treatment (day one, first sampling), 7 days using mouthwash, final sampling (day 8)
  Quantification of E. gingivalis DNA levels using quantitative polymerase chain reaction (qPCR) before (day 1) and after (day 8) using the mouthwash octenident® twice daily for seven days. Total DNA will be isolated from plaque and saliva samples on day 1 and day 8. The outcome will be reported as the absolute change in E. gingivalis DNA concentration from baseline to post-treatment. A standard curve will be generated using a dilution series of DNA with known concentrations. DNA concentrations in study samples will be interpolated from this curve to assess absolute changes in DNA quantity before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Koehsler, Prof. Dr., Principal Investigator — Institute for Specific Prophylaxis and Tropical Medicine, Medical University of Vienna
Locations (1):
- Institute for Specific Prophylaxis and Tropical Medicine, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
not relevant for this study

REFERENCES:
- [Background] Bonner M, Amard V, Bar-Pinatel C, Charpentier F, Chatard JM, Desmuyck Y, Ihler S, Rochet JP, Roux de La Tribouille V, Saladin L, Verdy M, Girones N, Fresno M, Santi-Rocca J. Detection of the amoeba Entamoeba gingivalis in periodontal pockets. Parasite. 2014;21:30. doi: 10.1051/parasite/2014029. Epub 2014 Jul 2. PMID 24983705
- [Background] Kung E, Pietrzak J, Klaus C, Walochnik J. In vitro effect of octenidine dihydrochloride against Trichomonas vaginalis. Int J Antimicrob Agents. 2016 Mar;47(3):232-4. doi: 10.1016/j.ijantimicag.2015.12.010. Epub 2016 Jan 21. PMID 26899578
- [Background] Kohsler M, Kniha E, Wagner A, Walochnik J. Pilot Study on the Prevalence of Entamoeba gingivalis in Austria-Detection of a New Genetic Variant. Microorganisms. 2023 Apr 22;11(5):1094. doi: 10.3390/microorganisms11051094. PMID 37317068